CLINICAL TRIAL: NCT00383006
Title: Affect Management Group for Adult Survivors of Childhood Trauma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulties in finding enough study participants.
Sponsor: University of Zurich (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSYUNIZH26092006
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Psychotherapy, Group; Stress Disorders, Post-Traumatic; Ambulatory Care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Skills for affect regulation (behavior)

SUMMARY:
Problems of self regulation, e.g. emotional dysfunction, represent a core symptom of adult patients with traumatic childhood experiences. The study intends to evaluate the efficiency of a 14-week group therapy for adult survivors of relational trauma in childhood. Main interventions are psychoeducation about the sequelae of childhood trauma, teaching of skills for affect regulation and techniques for activating resources. The hypothesis is that the group therapy significantly improves the participant's capacity in emotion management and self-soothing.

DETAILED DESCRIPTION:
Problems of self regulation, e.g. emotional dysfunction, represent a core symptom of adult patients with traumatic childhood experiences. Since sufficient capacity for self soothing and emotional regulation are essential for trauma exposure, modern trauma therapy concepts are phase-oriented, beginning with working on "stabilization". The study intends to evaluate the efficiency of a 14-week group therapy for adult survivors of relational trauma in childhood. Main interventions are psychoeducation about the sequelae of childhood trauma, teaching of skills for affect regulation and techniques for activating resources. Inclusion criteria are clinical significant problems with self-regulation and the presence of childhood trauma. Outcome measures are based on self-rating questionnaires, clinical interviews and an experimental computer-task at timepoint pre-, post- and 3-month-follow-up. There is no control condition in the pilot-study phase.

ELIGIBILITY:
Inclusion Criteria:

* Adults with moderate to severe relational trauma in childhood (emotional, sexual or physical abuse, emotional or physical neglect)
* DSM-IV diagnosis of posttraumatic stress disorder

Exclusion Criteria:

* Severe dissociation
* Environmental safety problems
* Ongoing enmeshment with perpetrators
* Psychotic disorders
* Severe depression
* Acute suicidality
* Substance abuse
* Severe cognitive decline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2006-05; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Score on affect regulation capacity at week 14(post-interventional) and month 3 (follow-up) | 2008

SECONDARY OUTCOMES:
Score on depression at week 14 (post-interventional) and month 3 (follow-up) | 2008
Score on life quality at week 14 (post-interventional) and month 3 (follow-up) | 2008
Score on personal resources at week 14 (post-interventional) and month 3 (follow-up) | 2008

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Mueller, MD, Principal Investigator — Department of Psychiatry, University Hospital, 8091 Zurich, Switzerland; Michael Rufer, MD, Principal Investigator — Department of Psychiatry, University Hospital, 8091 Zurich, Switzerland
Locations (1):
- Department of Psychiatry, University Hospital, Zurich, Canton of Zurich, Switzerland